CLINICAL TRIAL: NCT00172328
Title: Antibody Response and Immune Memory 15-18 Years After HBV Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 930306
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-09

CONDITIONS: Hepatitis B; Vaccine
Keywords: Hepatitis B; vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: Hepatitis B vaccine

SUMMARY:
Taiwan is an endemic region for hepatitis B. Before the implementation of a nationwide vaccination program in 1984, the hepatitis B virus (HBV) carrier rate in the general population was 15 to 20%.1-2 The major impact of hepatitis B (HB) infection is its long-term sequelae which may include chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma.3 Perinatal infection accounts for 40-50% of all hepatitis B infections and is responsible for the generation-to-generation transmission of HB virus.4 Hepatitis B vaccines, both plasma derived and recombinant, are highly immunogenic and efficacious.5-10 It has been reported that HB vaccine given soon after birth is able to protect infants from perinatal infection and HB infection became the first disease model to show that mother-to-neonate transmission can be interrupted by an effective vaccine.11 Taiwan started a national program of HB vaccination since 1984. This program resulted in a significant reduction of the HB carrier rate in children aged below 10 years from 9.8% before nationwide vaccination to 1.3% after the program.12 It also decreased the incidence of hepatocellular carcinoma in children aged 6 to 9 years from 0.52 to 0.13 per 100,000.13 However, the duration of protection provided by the HB vaccine and the proper timing of a booster dose remains unclear. Because the HB vaccine is a subunit protein vaccine, which contains only HBsAg, a limited duration of protection is anticipated. The results of several long-term follow-up studies of the protective efficacy of HB vaccination have been published. Soon after vaccination, protective levels of antibody (anti-HBs >10 mIU/mL) can be detected in the great majority (83-99%) of vaccinees.5-7 The proportion of vaccinees with protective anti-HBs levels decreases to 75-87% 5 years after vaccination and further drops to 50 to 70% 10-12 years after.10,11,14,15,19-21 Because of the progressive decline of anti-HBs and the associated increased likelihood of development of new HBV infections, some investigators advise the use of a booster vaccination.20,21 However, a preponderance of data indicates that the protective efficacy of the HB vaccine can last for at least 5 to 10 years and a booster before 5 years is not necessary.16-18,22,23 By demonstrating significant augmentation of cellular immunity and adequate induction of a protective level of antiHBs (>10 mIU/ml) in HBsAg and HBeAg-positive subjects 10 years after HB vaccination, we also proved that protection afforded by HB vaccination persisted for no less than 10 years in all vaccinees.R Nevertheless, the protective efficacy after the period of 10 years remains unknown. Knowledge of the duration of protection of HB vaccine and the optimal timing of booster vaccination remains crucial. In this study, we are going to examine the humoral and cellular immunity and monitored the antibody response following a booster dose of HB vaccine in a group of children whom had been vaccinated 14 years prior to this study.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years old healthy individuals

Exclusion Criteria:

* Unhealthy individuals and those who refuse to participate

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Lu CY, Chiang BL, Chi WK, Chang MH, Ni YH, Hsu HM, Twu SJ, Su IJ, Huang LM, Lee CY. Waning immunity to plasma-derived hepatitis B vaccine and the need for boosters 15 years after neonatal vaccination. Hepatology. 2004 Dec;40(6):1415-20. doi: 10.1002/hep.20490. PMID 15565627